CLINICAL TRIAL: NCT00001092
Title: The Determinants of the Biology of HIV Transmission to Determine the Immunologic and Virologic Characteristics of Those Who May Have Transmitted HIV to Another Individual
Brief Title: The Biology of HIV Transmission
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: AI-05-007; UCSD Project 98-0776; AEHIV 007; AIEDRP AI-05-007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infections
Keywords: Semen; HIV-1; Sexual Partners; Drug Resistance, Microbial; CD8-Positive T-Lymphocytes; Saliva; Blood; Cervix Uteri; Vagina; Acute Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, genital fluids, and saliva collection

SUMMARY:
The purpose of this study is to look at the amount of HIV in the blood, genital fluid, and saliva of the partners of patients with early HIV infection. This study will also look at the strength of the immune systems of patients with early HIV infection.

Because HIV multiplies very quickly in the early stages of infection, patients with early HIV infection may be more likely to transmit HIV to their partners. The amount of HIV in blood, genital fluid, and saliva may determine the risk for transmission.

DETAILED DESCRIPTION:
Persons with early HIV infection may represent high transmission risk to their partners. Early infection, characterized by rapid virologic replication, insufficient immunologic control of infection, and more rapid course of disease progression, may be associated with increased infectiousness. The viral determinants of transmission may in part be explained by viral burden in blood, genital fluids, and oral cavity fluids. All three fluids may be the source for transmitted virus.

Persons with suspected HIV infection are asked to identify their possible source partners. The importance of partner referral is emphasized and assisted recruitment or active tracing is offered if necessary. Source partners will not be approached uninvited. If a partner states that he/she does not want to be contacted, then he/she will not be contacted further for the purpose of this study or for any other study. All patients are offered HIV counseling and plasma testing for HIV-1 RNA and CD4+ cells. Blood specimens are collected for plasma determination, and cellular and plasma fractions are collected for CAF and neutralization antibodies. Neutralization assays are used to detect humoral immune response in patients with primary HIV infection. Genital fluids and saliva are analyzed for viral RNA. Patients are seen in the clinic on Day 1 for blood draw and return 2 weeks later for blood test results. A follow-up period of at least 4 weeks is planned. Compensation is provided to all patients.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Have sex with or share injection drugs with a person who is thought to have early HIV infection, or if they have recently become HIV-positive.
* Can provide written consent.
* Are available for a follow-up period of at least 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected adults with recent seroconversion
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 1999-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kahn, Principal Investigator; Margaret Chesney, Principal Investigator; Rick Hecht, Principal Investigator; Susan Little, Principal Investigator; Eric Daar, Principal Investigator; Jay Levy, Principal Investigator; Robert Grant, Principal Investigator
Locations (3):
- United States (3):
  - Cedars Sinai Med Ctr, Los Angeles, California
  - UCSD, San Diego, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California